CLINICAL TRIAL: NCT04773041
Title: Connectomic Analysis in Dementia With Lewy Bodies: A Potential Diagnostic Imaging Biomarker
Brief Title: Dementia With Lewy Bodies - Infinitome
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A21-037
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2023-10

CONDITIONS: Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with DLB: Patients diagnosed with DLB enrolled from the HealthPartners Neuroscience Center.
  Interventions: Procedure: Infinitome
- Patients with Alzheimer's disease (AD): Patients diagnosed with AD age and sex-matched, selected from the ADNI database.
  Interventions: Procedure: Infinitome
- Patients with normal cognition (CN): Patients diagnosed with normal cognition age and sex-matched, selected from the ADNI database.
  Interventions: Procedure: Infinitome

INTERVENTIONS:
Procedure: Infinitome — All patients will have rs-FMRI images analyzed with the Infinitome cloud-based software processing program.

SUMMARY:
Dementia with Lewy bodies (DLB) is the second most common cause of dementia and is associated with parkinsonism, hallucinations, and cognitive fluctuations. Diagnosis is often either missed or delayed due to physician lack of familiarity with characteristic features, the inability of structural MRI to detect a pathological signature for this condition, and the lack of healthcare provider access to "indicative biomarkers" that are either unavailable at community clinics or costly due to lack of insurance coverage. The role of resting state function MRI (rs-fMRI) as a diagnostic biomarker has been underexplored in this disease. We propose using a novel cloud-based automated imaging software processing program that identifies abnormal brain networks or connectomes using resting state functional MRI (rs-fMRI) and data from the Human Connectome Project (HCP). Furthermore, the imaging protocol to capture this data is relatively short (15 minutes) and can be performed at most imaging centers, lending potential clinical applicability to this study. We intend to study dysfunctional large scale brain networks (LSBNs) in DLB by comparing rs-fMRI imaging data in this population with cognitively normal (CN) and mild Alzheimer's disease (AD) subjects from the Alzheimer's Disease Neuroimaging Initiative (ADNI)-2/3 database.

DETAILED DESCRIPTION:
Omniscient, a for-profit, Sydney, Australia-based company, created the cloud-based software Infinitome, a program that utilizes data from the Human Connectome Project (HCP) together with machine learning to analyze diffusion tensor and resting-state fMRI imaging data from remote sites. The foundation for this imaging tool is based upon the HCP atlas, which has also informed prior publications from our group, including the Connectomic Atlas of the Human Cerebrum (Baker, Burks, Briggs, Conner, et al. 2018). The Infinitome program creates a subject specific version of the Human Connectome Project Multimodal Parcellation (HCP-MMP1) atlas using diffusion tractography. Analytics are performed on both diffusion tensor imaging and rs-fMRI. Outlier detection using a tangent space connectivity matrix is performed by comparing results with a subset of 300 normal HCP subject fMRI samples to determine the range of normal correlations for each regions of interest in a large scale brain network which include:

1. Locus coeruleus vs. Nucleus basalis of Meynert
2. Locus coeruelus vs. Intralaminar nucleus of the thalamus
3. Nucleus basalis of Meynert vs. Intralaminar nuclei of the thalamus
4. FST in the vs. Area PH in the lateral occipital lobe
5. Substantia nigra vs. Caudate nucleus Clinical Measures will be correlated with functional connectivity scores to identify relationship between clinical symptoms and large scale brain networks in DLB

ELIGIBILITY:
Inclusion Criteria:

* Age 40-90 years
* Established DLB diagnosis
* Mini mental status exam (MMSE) >15

Exclusion Criteria:

* Other forms of dementia including, but not limited to Alzheimer's dementia, frontotemporal dementia, vascular dementia, normal pressure hydrocephalus (NPH), etc,
* Inability to tolerate brain function magnetic resonance imaging (fMRI)
* Risk of brain fMRI due to implants or metal.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HealthPartners Neurology Clinic in Saint Paul, MN undergoing care for DLB and subjects included in the ADNI database.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Rosenbloom, MD, Principal Investigator — HealthPartners Neurology
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Alzheimer's Disease (AD): Patients diagnosed with AD age and MMSE-matched, selected from the ADNI database.
  Infinitome: All patients will have rs-FMRI images analyzed with the Infinitome cloud-based software processing program.
- Patients With Normal Cognition (CN): Patients diagnosed with normal cognition age matched, selected from the ADNI database.
  Infinitome: All patients will have rs-FMRI images analyzed with the Infinitome cloud-based software processing program.
Period: Overall Study
Arm/Group | Patients With DLB | Patients With Alzheimer's Disease (AD) | Patients With Normal Cognition (CN)
Started | 19 | 36 | 36
Completed | 18 | 36 | 36
Not Completed | 1 | 0 | 0
Not completed — Unable to data match | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Normal Cognition (CN): Patients diagnosed with normal cognition age-matched, selected from the ADNI database.
  Infinitome: All patients will have rs-FMRI images analyzed with the Infinitome cloud-based software processing program.
- Total: Total of all reporting groups
Arm/Group | Patients With DLB | Patients With Alzheimer's Disease (AD) | Patients With Normal Cognition (CN) | Total
Number analyzed (Participants) | 18 | 36 | 36 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (6.6) | 76 (7.3) | 74 (6.3) | 75 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 11 | 41
  Male | 3 | 21 | 25 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 4 | 5
  Not Hispanic or Latino | 18 | 35 | 32 | 85
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 6 | 8
  White | 18 | 32 | 29 | 79
  More than one race | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Education years [Mean (Standard Deviation); unit: years] | 17 (4) | 16 (3.6) | 16 (.99) | 16 (4.1)
Mini-Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The MMSE is a test that uses a series of questions to assess cognitive function. The total MMSE score was measured. Range: [0-30]. Higher score indicates better cognitive function.
  units on a scale | 23 (2.2) | 23 (2.6) | 29 (2.6) | 26 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Functional Connectivity Scores Between Pairs of Large Scale Brain Networks.
Description: Identify functional connectivity scores between pairs of large scale brain networks as determined by connectomic analysis using rs-fMRI Infinitome software in order to compare functional connectivity scores between groups. Eight parcellation pairs were chosen as primary pairs of interest.
  For each parcellation pair - Range [-1,1]. Higher positive score indicates greater connectivity.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: connectivity score
Arm/Group | Patients With DLB | Patients With Alzheimer's Disease (AD) | Patients With Normal Cognition (CN)
Number analyzed (Participants) | 18 | 36 | 36
connectivity score
  PH_right and FST_left | 0.164 (0.008) | 0.374 (0.006) | 0.344 (0.006)
  PH_right and FST_right | 0.340 (0.010) | 0.517 (0.006) | 0.442 (0.005)
  PH_all and FST_left | 0.307 (0.009) | 0.456 (0.006) | 0.433 (0.006)
  PH_all and FST_right | 0.359 (0.011) | 0.530 (0.005) | 0.493 (0.005)
  SubNigComp_left and Caud_left | 0.124 (0.012) | 0.122 (0.005) | 0.132 (0.004)
  SubNigComp_left and Caud_right | 0.134 (0.006) | 0.112 (0.005) | 0.144 (0.005)
  SubNigComp_right and Caud_left | 0.088 (0.012) | 0.127 (0.003) | 0.130 (0.004)
  SubNigComp_right and Caud_right | 0.063 (0.01) | 0.123 (0.004) | 0.123 (0.004)

2. Secondary Outcome: Correlation of Clinical Measures and Functional Connectivity Scores
Description: Clinical Measures will be correlated with functional connectivity scores to identify relationship between clinical symptoms and large scale brain networks in DLB . Range [-1,1]. Higher score indicates greater connectivity.
  Correlation of:
  1. Caudate R/Substantia Nigra R and Clock Drawing Test
  2. Caudate R/Substantia Nigra R and ADAS Number Cancellation
  3. PH R/FST R and ADAS Construction Praxis
  4. PH R/FST R and Clock Drawing Test
Time Frame: Baseline
Measure: Number; unit: correlation coefficient
Arm/Group | Patients With DLB | Patients With Alzheimer's Disease (AD) | Patients With Normal Cognition (CN)
Number analyzed (Participants) | 18 | 36 | 36
correlation coefficient
  Caudate R/Substantia Nigra R and Clock Drawing Test | -0.50 | -0.23 | 0.26
  Caudate R/Substantia Nigra R and ADAS Number Cancellation | -0.65 | -0.01 | -0.06
  PH R/FST R and ADAS Construction Praxis | -0.31 | -0.05 | -0.02
  PH R/FST R and Clock Drawing Test | -0.17 | 0.18 | -0.03

ADVERSE EVENTS:
Time Frame: 2 months for DLB patients, No adverse event data collected for AD or CN patients.
Description: Adverse event data was not collected for AD and CN patients - study data was from ADNI-2/3 database.
Arm/Group | Patients With DLB | Patients With Alzheimer's Disease (AD) | Patients With Normal Cognition (CN)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/18 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
DLB patients (n=18) were matched 2:1 to two control groups taken from the ADNI database: older adults with AD/CI confirmed by biomarkers and/or PET testing, and older adults who were cognitively normal with negative results from biomarker and/or PET testing. Both groups were matched by age, but only the AD/CI group was matched by MMSE score. Matching by sex was not possible due to the high prevalence of men in the DLB sample (83%) vs ADNI (46% male).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT04773041/Prot_SAP_000.pdf